CLINICAL TRIAL: NCT04754698
Title: Immunogenicity and Safety of the CoronaVac Vacccine in Patients With Autoimmune Rheumatic Diseases and People Living With HIV/AIDS
Brief Title: COVID-19 CoronaVac in Patients With Autoimmune Rheumatic Diseases and HIV/AIDS
Acronym: CoronavRheum
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 42566621.0.0000.0068
Record Dates: First submitted 2021-02-08; First posted 2021-02-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-11

CONDITIONS: Rheumatic Disease; HIV Infections; AIDS; Safety Issues; Immunogenicity; COVID-19
Keywords: CoronaVac; Vaccine; Rheumatic disease; Systemic lupus erythematosus; Rheumatoid arthritis; HIV; AIDS; Safety; Immunogenicity; COVID-19
MeSH Terms: conditions — Rheumatic Diseases; HIV Infections; Acquired Immunodeficiency Syndrome; COVID-19; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Study consisting of 3 arms, all of which will receive CoronaVac: patients with rheumatic diseases, PLWHA, and healthy controls. Also, in an exploratory, post hoc, substudy nested within the trial, 2 other arms will receive exercise or no intervention 1 hoour before the third dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with rheumatic diseases (Other): CoronaVac 2-dose schedule with 21-28-day interval and a booster dose (third dose of CoronaVac) 6 months after the primary vaccination
  Interventions: Biological: CoronaVac
- Patients with PLWHA (Other): CoronaVac 2-dose schedule with 21-28-day interval
  Interventions: Biological: CoronaVac
- Healthy controls (Other): CoronaVac 2-dose schedule with 21-28-day interval and a booster dose (third dose of CoronaVac) 6 months after the primary vaccination
  Interventions: Biological: CoronaVac

INTERVENTIONS:
Biological: CoronaVac — CoronaVac (Sinovac Biotech Ltd., Beijing, China)

SUMMARY:
Patients with chronic rheumatic diseases (such as systemic lupus erythematosus [SLE], rheumatoid arthritis [RA], ankylosing spondylitis [AS], juvenile idiopathic arthritis [JIA], poly/dermatomyositis [PM/DM], systemic sclerosis [SSc], systemic vasculitis, and primary Sjögren's syndrome [pSS]) are particularly susceptible to infectious diseases due to autoimmune disorder itself and its treatment (immunosuppressive therapies). Similarly, people living with HIV/AIDS (PLWHA) are predisposed to infections by different agents.

The current 2019 Coronavirus Disease Pandemic-19 (COVID-19), caused by the SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) began in December 2019 in Wuhan, China, and quickly became a global health and economic emergency by taking to an unprecedented burden on health systems around the world.

However, SARS-Cov-2 infection raised particular concern in patients with autoimmune rheumatic diseases (DRAI) since, due to chronic inflammatory immune dysregulation and the regular use of immunosuppressive drugs, these patients are considered to be at high risk of contracting SARS-CoV-2 and potentially evolving to a worse prognosis.

The overlap between the COVID-19 pandemic and the HIV/AIDS pandemic also poses an additional challenge, as the impact of co-infection is not yet fully known. The response to vaccines for other agents, however, has already been described as compromised in PLWHA.

Vaccination is the most effective preventive measure to control the spread of coronavirus and to reduce associated complications. Usually, live or attenuated vaccines are not recommended for patients with chronic rheumatic diseases using immunosuppressants. However, immunization with inactivated agents is strongly indicated, resulting, in general, in good immunogenicity and adequate vaccine safety, as well as without relevant deleterious effects on diseases.

Vaccine efficacy studies are needed to verify the immunogenicity of the vaccine against COVID-19 in immunosuppressed patients with rheumatological disease and those with HIV-related disease considering the risk of greater severity. In addition, it is important to assess the safety of the vaccine in this population as well as the possibility of reactivating the rheumatological disease itself.

The present study will evaluate the safety and immunogenicity of the CoronaVac (Coronavirus vaccine, Sinovac Biotech Ltd.) in patients with rheumatic diseases and PLWHA

DETAILED DESCRIPTION:
A sample of 1254 patients with rheumatic diseases and 542 healthy controls matched for age and sex was calculated as follows.

1.A) Evaluation of patients with SLE compared to a healthy control group matched for age and sex. The investigators calculated 74 patients in each arm, which will be compared independently to the healthy control group:

* 74 SLE patients treated with hydroxychloroquine alone;
* 74 SLE patients with mild immunosuppression (azathioprine or methotrexate and prednisone <10 mg/day);
* 74 patients with moderate to severe immunosuppression (mycophenolate mofetil or cyclophosphamide and/or prednisone >10 mg/day);
* 50 patients with belimumab (convenience sample). Total: 272 SLE patients and 74 healthy controls.

  1.B) Evaluation of RA patients compared to healthy controls matched for age and sex. The investigators calculated 61 patients in each arm, which will be independently compared to the control group:
* 61 RA patients only with conventional synthetic disease-modifying drugs (DMARDs);
* 61 RA patients with biological disease-modifying drugs (bDMARDs) with anti-TNF (anti-tumor necrosis factor) action;
* 61 RA patients with bDMARDs with non-anti-TNF action and with impact on the production of immunoglobulins (abatacept and rituximab);
* 61 RA patients with bDMARDs with anti-IL-6 (anti-interleukin-6) action (tocilizumab) and synthetic drugs with anti-JAK (anti-janus kinase) action (tofacitinib).

Total: 244 RA patients vs. 61 healthy controls. 1.C) Evaluation of the interruption of the use of methotrexate (MTX) for 4 weeks from the first dose of vaccination in RA patients. Inclusion: patients using MTX in a stable dose for at least 4 weeks, prednisone maximum dose of 7.5 mg/day, in association or not with other drugs, to be randomized in two arms: one that keeps the therapy stable and the other which suspends MTX for 4 weeks from the first dose. The investigators calculated 96 patients in each arm:

* 96 MTX patients who will not have their therapy changed;
* 96 MTX patients who will stop only MTX on the day of vaccination for 4 weekly applications.

Total: 192 RA patients.

1.D) Evaluation of patients with AS/psoriatic arthritis compared to a healthy control group matched for age and sex. The investigators calculated 136 patients in each arm, 136 with synthetic DMARDs and 136 with bDMARDs, to be compared with 136 healthy controls matched for age and sex.

Total: 272 patients with AS/psoriatic arthritis vs. 136 healthy controls.

1. E) A convenience sample of 250 (50 in each group) patients with other rare rheumatic diseases (SSc, PM/DM, pSS, systemic vasculitis, and primary antiphospholipid antibody syndrome) being followed up in Rheumatology Division (HCFMUSP) will be vaccinated and matched using the pool of controls from the other samples.

   Controls: 271 healthy controls matched for age and sex will be included according to the need for controls for SLE (n = 74), RA (n = 61) and AS/psoriatic arthritis (n = 136) will be selected to receive the vaccine at HCFMUSP.
2. PEOPLE LIVING WITH HIV/AIDS (PLWHA) The investigators considered the immunogenicity of the vaccine for Yellow Fever as a parameter in a previous study carried out by our group. The response found was p1 = 92% induction of neutralizing antibodies in PLWHA. Considering the 1:1 ratio between vaccinated and controls, alpha error of 5% with 80% power, the sample size will be 271 vaccinated in the PLWHA group and 271 in the control group, with an effect size of 0.25.

Total population: 1254 ARD patients + 542 controls + 271 patients in PLWHA group = 2067 patients.

In addition to a symptom diary (provided to research subjects on the 1st and 2nd vaccine doses), all patients and controls were instructed to contact the researchers by email, WhatsApp, and telephone in case of adverse effects or symptoms of COVID. In cases of suspected COVID, RT-PCR and genotyping are being performed.

Extension phase of the project

There are clinical trials using a booster dose (third dose of mRNA vaccine against COVID-19) in renal transplant recipients, who similarly to patients with autoimmune rheumatic diseases (ARDs), had high rates (about 40%) of poor humoral response. Antibody titers increased after the third dose in one third of patients who had negative response and in all patients who had low antibody titers. In addition, patients on therapy with specific drugs (tacrolimus, mycophenolate and glucocorticoids) were less likely to develop anti-SARS-CoV-2 antibodies than those treated with other regimes. No serious adverse events were observed after the third dose (Werbel et al., 2021; Benotmane et al., 2021).

Therefore, we consider a booster dose (third dose of Sinovac-CoronaVac) for ARDs patients 6 months after the primary vaccination. The monitoring of anti-SARS-CoV-2 humoral response [anti-SARS-CoV-2 IgG seroconversion and neutralizing antibody (NAb)] will be carried out immediately before the third dose and 6 weeks after.

This extension phase of the study was approved by the National Research Ethics Committee (Comissão Nacional de Ética em Pesquisa) (4.951.263). Only participants (patients/controls) who agree to participate in the extension phase of the study will be included according to the signed updated informed consent form. The expected sample is 1300 patients and 340 controls.

Guidance on use of immunosuppressive medications during the vaccination period will be according to the updated recommendations of the American College of Rheumatology (ACR) (https://www.rheumatology.org/Portals/0/Files/COVID-19-Vaccine-Clinical-Guidance-RheumaticDiseasesSummary.pdf).

Similar to the first phase of the study, in addition to a symptom diary (provided to research subjects on the 3th vaccine doses), all patients and controls were instructed to contact the researchers by email, WhatsApp, and telephone in case of adverse effects or symptoms of COVID. In cases of suspected COVID, RT-PCR and genotyping are being performed.

In an exploratory substudy nested within this phase 4 trial, a subsample composed by AS/psoriatic arthritis (n=60) will be randomly assigned to receive exercise or nothing 1 hour before vaccination, under the working hypothesis that exercise may boost immune responses to the vaccine, wich would benefit immunocompromised patients. The exercise session will be conducted by experienced exercise physiologists and will comprise a brief specific warm-up and 3 unilateral resistance exercises (lateral raise, biceps curl and overhead extension) in the left arm (the same arm used for vaccination). The exercises will be performed using dumbbells, with eccentric and concentric contractions (4 sets of 8-12 repetition maximum). Interval between exercises and sets will be 30 seconds. The total duration of the exercise session will be approximately 20 minutes. Thirty minutes after the end of the exercise session, patients will receive the vaccine in the same arm (i.e., left arm). Immediately, 24h and 48h after the exercise session, local pain (muscle soreness) in the exercised arm will be assessed by visual analogue scale (0 [no pain] to 100 [worst possible pain]). Exercise-induced edema will be determined by circumference measures of the biceps. Participants will also report self-perceived exertion after exercise using the Borg scale. Blood sample to assess immunogenicity (primary outcome) will follow the same schedule proposed in the phase 4 trial. Control group will receive no intervention and will follow the vaccination scheme adopted in the phase 4 trial.

Amendment to the extension phase of the project

Rationale: There are clinical trials comparing homologous vaccine scheme (two first doses) against COVID-19 versus heterologous immunization suggesting that the latter was well tolerated and improved immunogenicity healthy individuals (Hillus et al., 2021). In animal models, there is evidence that application of a third vaccine dose (booster) with an mRNA vaccine after two vaccine doses of inactivated against COVID-19 induce a relatively higher level of neutralizing antibodies and T cell response (Zhang et al., 2021). Thus, we will include the following extension analyses in this project:

1. For patients and controls without humoral response (anti-SARS-CoV-2 S1/S2 IgG and/or neutralizing antibodies) after the 3rd dose of CoronaVac vaccine, a booster dose with the available heterologous vaccine will be given as per the Plan National Vaccination of COVID-19 in ARD patients.
2. A new serology analysis will be performed (anti-SARS-CoV-2 S1/S2 IgG and neutralizing antibodies) 4-8 weeks after the heterologous vaccine booster. Immunogenicity will be assessed through seroconversion rates of total IgG antibodies against S1 and S2 antigens and neutralizing antibodies.
3. In addition, the participants will be instructed to write down in a diary standardized changes that occur and to contact investigators by e-mail or WhatsApp.
4. The updated recommendations of the American College of Rheumatology (ACR) regarding to the use of immunosuppressive medications during the vaccination period will be followed (https://www.rheumatology.org/Portals/0/Files/COVID-19-Vaccine-Clinical-Guidance-RheumaticDiseasesSummary.pdf).

This amendment to the extension phase of the project was approved by the National Research Ethics Committee (Comissão Nacional de Ética em Pesquisa) (5.014.175). Only participants (patients/controls) who agree to participate in this amendment to extension phase of the study will be included according to the signed updated informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* RA patients according to the classification criteria of the European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR).
* Patients with axial spondyloarthritis (ASAS criteria 2009) and psoriatic arthritis (CASPAR 2012 criteria).
* SLE patients according to the SLICC classification criteria.
* SSc patients according to the ACR preliminary criteria.
* Patients with inflammatory myopathies according to the Bohan and Peter's criteria.
* Patients with primary vasculitis.
* Patients with pSS (2002 American-European Consensus group criteria and/or 2016 classification criteria of the EULAR/ACR.
* Patients with primary APS (primary antiphospholipid syndrome) (Sydney classification criteria).
* Patients with HIV-related illness.

Exclusion Criteria:

* History of anaphylactic response to vaccine components.
* Acute febrile illness.
* Guillain-Barré syndrome, decompensated heart failure (class III or IV), demyelinating disease.
* History of live virus vaccine up to 4 weeks before, virus vaccine inactivated up to 2 weeks before.
* History of having received blood products up to 6 months before the study.
* Individuals who do not accept to participate in the study and/or whose guardians do not agree to participate in the study.
* Hospitalized patients.
* Patients with severe conditions requiring hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2196 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Immunogenicity 1 | 8 months
  Presence of ≥30% of neutralizing activity of SARS-CoV-2 antibodies
Immunogenicity 2 | 8 months
  Seroconversion rate of anti-SARS-Cov-2 IgG antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Kallas, MD, PhD, Study Chair — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arend WP, Michel BA, Bloch DA, Hunder GG, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Takayasu arteritis. Arthritis Rheum. 1990 Aug;33(8):1129-34. doi: 10.1002/art.1780330811. PMID 1975175
- [Background] Avelino-Silva VI, Miyaji KT, Hunt PW, Huang Y, Simoes M, Lima SB, Freire MS, Caiaffa-Filho HH, Hong MA, Costa DA, Dias JZ, Cerqueira NB, Nishiya AS, Sabino EC, Sartori AM, Kallas EG. CD4/CD8 Ratio and KT Ratio Predict Yellow Fever Vaccine Immunogenicity in HIV-Infected Patients. PLoS Negl Trop Dis. 2016 Dec 12;10(12):e0005219. doi: 10.1371/journal.pntd.0005219. eCollection 2016 Dec. PMID 27941965
- [Background] Avelino-Silva VI, Miyaji KT, Mathias A, Costa DA, de Carvalho Dias JZ, Lima SB, Simoes M, Freire MS, Caiaffa-Filho HH, Hong MA, Lopes MH, Sartori AM, Kallas EG. CD4/CD8 Ratio Predicts Yellow Fever Vaccine-Induced Antibody Titers in Virologically Suppressed HIV-Infected Patients. J Acquir Immune Defic Syndr. 2016 Feb 1;71(2):189-95. doi: 10.1097/QAI.0000000000000845. PMID 26361176
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (first of two parts). N Engl J Med. 1975 Feb 13;292(7):344-7. doi: 10.1056/NEJM197502132920706. No abstract available. PMID 1090839
- [Background] Brown LB, Spinelli MA, Gandhi M. The interplay between HIV and COVID-19: summary of the data and responses to date. Curr Opin HIV AIDS. 2021 Jan;16(1):63-73. doi: 10.1097/COH.0000000000000659. PMID 33186229
- [Background] Dougados M, van der Linden S, Juhlin R, Huitfeldt B, Amor B, Calin A, Cats A, Dijkmans B, Olivieri I, Pasero G, et al. The European Spondylarthropathy Study Group preliminary criteria for the classification of spondylarthropathy. Arthritis Rheum. 1991 Oct;34(10):1218-27. doi: 10.1002/art.1780341003. PMID 1930310
- [Background] Emmi G, Bettiol A, Mattioli I, Silvestri E, Di Scala G, Urban ML, Vaglio A, Prisco D. SARS-CoV-2 infection among patients with systemic autoimmune diseases. Autoimmun Rev. 2020 Jul;19(7):102575. doi: 10.1016/j.autrev.2020.102575. Epub 2020 May 5. PMID 32376395
- [Background] Fernandez-Ruiz R, Masson M, Kim MY, Myers B, Haberman RH, Castillo R, Scher JU, Guttmann A, Carlucci PM, Deonaraine KK, Golpanian M, Robins K, Chang M, Belmont HM, Buyon JP, Blazer AD, Saxena A, Izmirly PM; NYU WARCOV Investigators. Leveraging the United States Epicenter to Provide Insights on COVID-19 in Patients With Systemic Lupus Erythematosus. Arthritis Rheumatol. 2020 Dec;72(12):1971-1980. doi: 10.1002/art.41450. Epub 2020 Oct 28. PMID 32715660
- [Background] Furer V, Rondaan C, Heijstek MW, Agmon-Levin N, van Assen S, Bijl M, Breedveld FC, D'Amelio R, Dougados M, Kapetanovic MC, van Laar JM, de Thurah A, Landewe RB, Molto A, Muller-Ladner U, Schreiber K, Smolar L, Walker J, Warnatz K, Wulffraat NM, Elkayam O. 2019 update of EULAR recommendations for vaccination in adult patients with autoimmune inflammatory rheumatic diseases. Ann Rheum Dis. 2020 Jan;79(1):39-52. doi: 10.1136/annrheumdis-2019-215882. Epub 2019 Aug 14. PMID 31413005
- [Background] Garcia LF. Immune Response, Inflammation, and the Clinical Spectrum of COVID-19. Front Immunol. 2020 Jun 16;11:1441. doi: 10.3389/fimmu.2020.01441. eCollection 2020. PMID 32612615
- [Background] Gianfrancesco M, Hyrich KL, Al-Adely S, Carmona L, Danila MI, Gossec L, Izadi Z, Jacobsohn L, Katz P, Lawson-Tovey S, Mateus EF, Rush S, Schmajuk G, Simard J, Strangfeld A, Trupin L, Wysham KD, Bhana S, Costello W, Grainger R, Hausmann JS, Liew JW, Sirotich E, Sufka P, Wallace ZS, Yazdany J, Machado PM, Robinson PC; COVID-19 Global Rheumatology Alliance. Characteristics associated with hospitalisation for COVID-19 in people with rheumatic disease: data from the COVID-19 Global Rheumatology Alliance physician-reported registry. Ann Rheum Dis. 2020 Jul;79(7):859-866. doi: 10.1136/annrheumdis-2020-217871. Epub 2020 May 29. PMID 32471903
- [Background] Leavitt RY, Fauci AS, Bloch DA, Michel BA, Hunder GG, Arend WP, Calabrese LH, Fries JF, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Wegener's granulomatosis. Arthritis Rheum. 1990 Aug;33(8):1101-7. doi: 10.1002/art.1780330807. PMID 2202308
- [Background] Lightfoot RW Jr, Michel BA, Bloch DA, Hunder GG, Zvaifler NJ, McShane DJ, Arend WP, Calabrese LH, Leavitt RY, Lie JT, et al. The American College of Rheumatology 1990 criteria for the classification of polyarteritis nodosa. Arthritis Rheum. 1990 Aug;33(8):1088-93. doi: 10.1002/art.1780330805. PMID 1975174
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Ye C, Cai S, Shen G, Guan H, Zhou L, Hu Y, Tu W, Chen Y, Yu Y, Wu X, Chen Y, Zhong J, Dong L. Clinical features of rheumatic patients infected with COVID-19 in Wuhan, China. Ann Rheum Dis. 2020 Aug;79(8):1007-1013. doi: 10.1136/annrheumdis-2020-217627. Epub 2020 May 22. PMID 32444415
- [Background] Zhang Y, Zeng G, Pan H, Li C, Hu Y, Chu K, Han W, Chen Z, Tang R, Yin W, Chen X, Hu Y, Liu X, Jiang C, Li J, Yang M, Song Y, Wang X, Gao Q, Zhu F. Safety, tolerability, and immunogenicity of an inactivated SARS-CoV-2 vaccine in healthy adults aged 18-59 years: a randomised, double-blind, placebo-controlled, phase 1/2 clinical trial. Lancet Infect Dis. 2021 Feb;21(2):181-192. doi: 10.1016/S1473-3099(20)30843-4. Epub 2020 Nov 17. PMID 33217362
- [Background] Miyakis S, Lockshin MD, Atsumi T, Branch DW, Brey RL, Cervera R, Derksen RH, DE Groot PG, Koike T, Meroni PL, Reber G, Shoenfeld Y, Tincani A, Vlachoyiannopoulos PG, Krilis SA. International consensus statement on an update of the classification criteria for definite antiphospholipid syndrome (APS). J Thromb Haemost. 2006 Feb;4(2):295-306. doi: 10.1111/j.1538-7836.2006.01753.x. PMID 16420554
- [Background] Rudwaleit M, Landewe R, van der Heijde D, Listing J, Brandt J, Braun J, Burgos-Vargas R, Collantes-Estevez E, Davis J, Dijkmans B, Dougados M, Emery P, van der Horst-Bruinsma IE, Inman R, Khan MA, Leirisalo-Repo M, van der Linden S, Maksymowych WP, Mielants H, Olivieri I, Sturrock R, de Vlam K, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part I): classification of paper patients by expert opinion including uncertainty appraisal. Ann Rheum Dis. 2009 Jun;68(6):770-6. doi: 10.1136/ard.2009.108217. Epub 2009 Mar 17. PMID 19297345
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Tillett W, Costa L, Jadon D, Wallis D, Cavill C, McHugh J, Korendowych E, McHugh N. The ClASsification for Psoriatic ARthritis (CASPAR) criteria--a retrospective feasibility, sensitivity, and specificity study. J Rheumatol. 2012 Jan;39(1):154-6. doi: 10.3899/jrheum.110845. Epub 2011 Nov 15. PMID 22089469
- [Background] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism classification criteria for primary Sjogren's syndrome: A consensus and data-driven methodology involving three international patient cohorts. Ann Rheum Dis. 2017 Jan;76(1):9-16. doi: 10.1136/annrheumdis-2016-210571. Epub 2016 Oct 26. PMID 27789466
- [Background] Hillus D, Schwarz T, Tober-Lau P, Vanshylla K, Hastor H, Thibeault C, Jentzsch S, Helbig ET, Lippert LJ, Tscheak P, Schmidt ML, Riege J, Solarek A, von Kalle C, Dang-Heine C, Gruell H, Kopankiewicz P, Suttorp N, Drosten C, Bias H, Seybold J; EICOV/COVIM Study Group; Klein F, Kurth F, Corman VM, Sander LE. Safety, reactogenicity, and immunogenicity of homologous and heterologous prime-boost immunisation with ChAdOx1 nCoV-19 and BNT162b2: a prospective cohort study. Lancet Respir Med. 2021 Nov;9(11):1255-1265. doi: 10.1016/S2213-2600(21)00357-X. Epub 2021 Aug 13. PMID 34391547
- [Background] Zhang J, He Q, An C, Mao Q, Gao F, Bian L, Wu X, Wang Q, Liu P, Song L, Huo Y, Liu S, Yan X, Yang J, Cui B, Li C, Wang J, Liang Z, Xu M. Boosting with heterologous vaccines effectively improves protective immune responses of the inactivated SARS-CoV-2 vaccine. Emerg Microbes Infect. 2021 Dec;10(1):1598-1608. doi: 10.1080/22221751.2021.1957401. PMID 34278956
- [Derived] Silva CA, de Vinci Kanda Kupa L, Medeiros-Ribeiro AC, Pasoto SG, Saad CGS, Yuki EFN, Landim JIVD, Leda VHFE, de Camargo Correia LS, Sartori AF, Martins CCMF, Ribeiro CT, Waridel F, de Oliveira Martins VA, Shinjo SK, Andrade DCO, Sampaio-Barros PD, Neto EFB, Aikawa NE, Bonfa E. Post-acute COVID-19 in three doses vaccinated autoimmune rheumatic diseases patients: frequency and pattern of this condition. Adv Rheumatol. 2023 Jun 8;63(1):26. doi: 10.1186/s42358-023-00309-z. PMID 37291679
- [Derived] Pereira RMR, Dagostin MA, Caparbo VF, Sales LP, Pasoto SG, Silva CA, Yuki EFN, Saad CGS, Medeiros-Ribeiro AC, Kupa LVK, Fusco SRG, Martins VAO, Martins CCMF, Barbas CV, Shinjo SK, Aikawa NE, Bonfa E. Anti-SARS-CoV-2 inactivated vaccine in patients with ANCA-associated vasculitis: Immunogenicity, safety, antibody decay and the booster dose. Clinics (Sao Paulo). 2022 Nov 29;78:100150. doi: 10.1016/j.clinsp.2022.100150. eCollection 2023. PMID 36529052
- [Derived] Silva CA, Medeiros-Ribeiro AC, Kupa LVK, Yuki EFN, Pasoto SG, Saad CGS, Fusco SRG, Pereira RMR, Shinjo SK, Halpern ASR, Borba EF, Souza FHC, Guedes LKN, Miossi R, Bonfiglioli KR, Domiciano DS, Shimabuco AY, Andrade DCO, Seguro LPC, Fuller R, Sampaio-Barros PD, Assad APL, Moraes JCB, Goldenstein-Schainberg C, Giardini HAM, Silva HC, Martins VAO, Villamarin LEB, Novellino RS, Sales LP, Araujo CSR, Silva MSR, Filho DMN, Lopes MH, Duarte AJS, Kallas EG, Aikawa NE, Bonfa E. Immunogenicity decay and case incidence six months post Sinovac-CoronaVac vaccine in autoimmune rheumatic diseases patients. Nat Commun. 2022 Oct 3;13(1):5801. doi: 10.1038/s41467-022-33042-0. PMID 36192386
- [Derived] G S Saad C, S R Silva M, Sampaio-Barros PD, C B Moraes J, G Schainberg C, Goncalves CR, Shimabuco AY, Aikawa NE, F N Yuki E, G Pasoto S, V K Kupa L, K Aoyama R, S R Araujo C, Silva CA, Medeiros-Ribeiro AC, Bonfa E. Interaction of TNFi and conventional synthetic DMARD in SARS-CoV-2 vaccine response in axial spondyloarthritis and psoriatic arthritis. Joint Bone Spine. 2023 Jan;90(1):105464. doi: 10.1016/j.jbspin.2022.105464. Epub 2022 Sep 20. PMID 36150668
- [Derived] Gualano B, Lemes IR, da Silva RP, Pinto AJ, Mazzolani BC, Smaira FI, Sieczkowska SM, Aikawa NE, Pasoto S, Medeiros-Ribeiro AC, Saad C, Yuk E, Silva C, Swinton P, Hallal PC, Roschel H, Bonfa E. Physical activity and antibody persistence 6 months after the second dose of CoronaVac in immunocompromised patients. Scand J Med Sci Sports. 2022 Oct;32(10):1510-1515. doi: 10.1111/sms.14213. Epub 2022 Jul 26. PMID 35844042
- [Derived] Aikawa NE, Kupa LVK, Silva CA, Saad CGS, Pasoto SG, Yuki EFN, Fusco SRG, Shinjo SK, Andrade DCO, Sampaio-Barros PD, Pereira RMR, Chasin ACS, Shimabuco AY, Luppino-Assad AP, Leon EP, Lopes MH, Antonangelo L, Medeiros-Ribeiro AC, Bonfa E. Strong response after fourth dose of mRNA COVID-19 vaccine in autoimmune rheumatic diseases patients with poor response to inactivated vaccine. Rheumatology (Oxford). 2022 Dec 23;62(1):480-485. doi: 10.1093/rheumatology/keac301. PMID 35639644
- [Derived] Pasoto SG, Halpern ASR, Guedes LKN, Ribeiro ACM, Yuki ENF, Saad CGS, da Silva CAA, de Vinci Kanda Kupa L, Villamarin LEB, de Oliveira Martins VA, Martins CCMF, Deveza GBH, Leon EP, Bueno C, Pedrosa TN, Santos REB, Soares R, Aikawa NE, Bonfa E. Inactivated SARS-CoV-2 vaccine in primary Sjogren's syndrome: humoral response, safety, and effects on disease activity. Clin Rheumatol. 2022 Jul;41(7):2079-2089. doi: 10.1007/s10067-022-06134-x. Epub 2022 Mar 19. PMID 35306594
- [Derived] Aikawa NE, Kupa LVK, Medeiros-Ribeiro AC, Saad CGS, Yuki EFN, Pasoto SG, Rojo PT, Pereira RMR, Shinjo SK, Sampaio-Barros PD, Andrade DCO, Halpern ASR, Fuller R, Souza FHC, Guedes LKN, Assad APL, Moraes JCB, Lopes MRU, Martins VAO, Betancourt L, Ribeiro CT, Sales LP, Bertoglio IM, Bonoldi VLN, Mello RLP, Balbi GGM, Sartori AMC, Antonangelo L, Silva CA, Bonfa E. Increment of immunogenicity after third dose of a homologous inactivated SARS-CoV-2 vaccine in a large population of patients with autoimmune rheumatic diseases. Ann Rheum Dis. 2022 Jul;81(7):1036-1043. doi: 10.1136/annrheumdis-2021-222096. Epub 2022 Mar 11. PMID 35277389
- [Derived] Araujo CSR, Medeiros-Ribeiro AC, Saad CGS, Bonfiglioli KR, Domiciano DS, Shimabuco AY, Silva MSR, Yuki EFN, Pasoto SG, Pedrosa T, Kupa LVK, Zou G, Pereira RMR, Silva CA, Aikawa NE, Bonfa E. Two-week methotrexate discontinuation in patients with rheumatoid arthritis vaccinated with inactivated SARS-CoV-2 vaccine: a randomised clinical trial. Ann Rheum Dis. 2022 Jun;81(6):889-897. doi: 10.1136/annrheumdis-2021-221916. Epub 2022 Feb 22. PMID 35193873
- [Derived] Medeiros-Ribeiro AC, Bonfiglioli KR, Domiciano DS, Shimabuco AY, da Silva HC, Saad CGS, Yuki EFN, Pasoto SG, Araujo CSR, Nakai TL, Silva CA, Pedrosa T, Kupa LVK, Silva MSR, Balbi GGM, Kallas EG, Aikawa NE, Bonfa E. Distinct impact of DMARD combination and monotherapy in immunogenicity of an inactivated SARS-CoV-2 vaccine in rheumatoid arthritis. Ann Rheum Dis. 2022 May;81(5):710-719. doi: 10.1136/annrheumdis-2021-221735. Epub 2022 Feb 8. PMID 35135832
- [Derived] Gualano B, Lemes IR, Silva RP, Pinto AJ, Mazzolani BC, Smaira FI, Sieczkowska SM, Aikawa NE, Pasoto SG, Medeiros-Ribeiro AC, Saad CGS, Yuki EFN, Silva CA, Swinton P, Hallal PC, Roschel H, Bonfa E. Association between physical activity and immunogenicity of an inactivated virus vaccine against SARS-CoV-2 in patients with autoimmune rheumatic diseases. Brain Behav Immun. 2022 Mar;101:49-56. doi: 10.1016/j.bbi.2021.12.016. Epub 2021 Dec 23. PMID 34954325
- [Derived] Aikawa NE, Kupa LVK, Pasoto SG, Medeiros-Ribeiro AC, Yuki EFN, Saad CGS, Pedrosa T, Fuller R, Shinjo SK, Sampaio-Barros PD, Andrade DCO, Pereira RMR, Seguro LPC, Valim JML, Waridel F, Sartori AMC, Duarte AJS, Antonangelo L, Sabino EC, Menezes PR, Kallas EG, Silva CA, Bonfa E. Immunogenicity and safety of two doses of the CoronaVac SARS-CoV-2 vaccine in SARS-CoV-2 seropositive and seronegative patients with autoimmune rheumatic diseases in Brazil: a subgroup analysis of a phase 4 prospective study. Lancet Rheumatol. 2022 Feb;4(2):e113-e124. doi: 10.1016/S2665-9913(21)00327-1. Epub 2021 Dec 3. PMID 34901885
- [Derived] Sampaio-Barros PD, Medeiros-Ribeiro AC, Luppino-Assad AP, Miossi R, da Silva HC, Yuki EFVN, Pasoto SG, Saad CGS, Silva CA, Kupa LVK, Deveza GBH, Pedrosa TN, Aikawa NE, Bonfa E. SARS-CoV-2 vaccine in patients with systemic sclerosis: impact of disease subtype and therapy. Rheumatology (Oxford). 2022 Jun 28;61(SI2):SI169-SI174. doi: 10.1093/rheumatology/keab886. PMID 34894235
- [Derived] Yuki EFN, Borba EF, Pasoto SG, Seguro LP, Lopes M, Saad CGS, Medeiros-Ribeiro AC, Silva CA, de Andrade DCO, Kupa LVK, Betancourt L, Bertoglio I, Valim J, Hoff C, Formiga FFC, Pedrosa T, Kallas EG, Aikawa NE, Bonfa E. Impact of Distinct Therapies on Antibody Response to SARS-CoV-2 Vaccine in Systemic Lupus Erythematosus. Arthritis Care Res (Hoboken). 2022 Apr;74(4):562-571. doi: 10.1002/acr.24824. Epub 2022 Mar 4. PMID 34806342
- [Derived] Shinjo SK, de Souza FHC, Borges IBP, Dos Santos AM, Miossi R, Misse RG, Medeiros-Ribeiro AC, Saad CGS, Yuki EFN, Pasoto SG, Kupa LVK, Ceneviva C, Seraphim JC, Pedrosa TN, Vendramini MBG, Silva CA, Aikawa NE, Bonfa E. Systemic autoimmune myopathies: a prospective phase 4 controlled trial of an inactivated virus vaccine against SARS-CoV-2. Rheumatology (Oxford). 2022 Aug 3;61(8):3351-3361. doi: 10.1093/rheumatology/keab773. PMID 34664616
- [Derived] Medeiros-Ribeiro AC, Aikawa NE, Saad CGS, Yuki EFN, Pedrosa T, Fusco SRG, Rojo PT, Pereira RMR, Shinjo SK, Andrade DCO, Sampaio-Barros PD, Ribeiro CT, Deveza GBH, Martins VAO, Silva CA, Lopes MH, Duarte AJS, Antonangelo L, Sabino EC, Kallas EG, Pasoto SG, Bonfa E. Immunogenicity and safety of the CoronaVac inactivated vaccine in patients with autoimmune rheumatic diseases: a phase 4 trial. Nat Med. 2021 Oct;27(10):1744-1751. doi: 10.1038/s41591-021-01469-5. Epub 2021 Jul 30. PMID 34331051